CLINICAL TRIAL: NCT04370951
Title: Efficacy of the Erector Spinae Plane (ESP) Block for Quality of Recovery in Posterior Thoraco-Lumbar Spinal Decompression Surgery: A Randomised Control Trial
Brief Title: Efficacy of the Erector Spinae Plane Block in Posterior Thoraco- Lumbar Spinal Decompression Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Dylan Finnerty, Clinical Lecturer in Anaesthesia, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1/378/2088
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Spinal Surgery
Keywords: erector spinae plane block; post operative recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Patients will receive a ESP block with 20mls 0.25% Levobupivicaine bilaterally, pre incision plus standardised multimodal analgesia
  Interventions: Procedure: Erector Spinae Plane Block - Ultrasound guided
- Control (No Intervention): no ESP block, standardised multimodal analgesia

INTERVENTIONS:
Procedure: Erector Spinae Plane Block - Ultrasound guided — 20mls 0.25% Levobupivicaine ultrasound guided bilaterally
  Arms: Erector Spinae Plane Block

SUMMARY:
Spinal Surgery can be associated with significant post operative pain. This can be a considerable source of morbidity, resulting in a longer duration of in- hospital stay and increasing opiate requirements. As a result the patient experiences a more arduous recovery process.

Recently a new form of Regional Anaesthesia has been described for patients undergoing Spinal surgery. The Erector Spinae Plane Block involves depositing Local Anaesthetic under Ultra Sound guidance on top of the Transverse Process of the Spine and deep to the Erector Spinae Muscle. Patients who have had this procedure report lower pain scores and have a lesser opiate requirement in the post operative period.

DETAILED DESCRIPTION:
This study will test the hypothesis that patients receiving ESP Block have higher QoR-15 scores and better post operative analgesia in comparison with patients receiving standard care after Spinal Surgery.

Objectives & endpoints / outcome measures

1. The Primary outcome in this study will be the patient centred QoR-15 score among ESB and Control patients;
2. Secondary outcomes will be:

   1. Area under the VRS pain score versus time (24 hr post-op);
   2. VRS pain scores at 1 hr, 4 hr, 12 hr, 24 hr postop;
   3. time to administration of first rescue analgesia after the block;
   4. documentation of adverse events : hypotension, pruritus, nausea and vomiting
   5. DAH -30 Days at home at 30 Days

      Proposed sample size The established minimum clinically important difference in QoR-15 is 8.0 and the SD of QoR-15 scores after major surgery is in the order of 10 [range of QoR score is 1-150]. Therefore, assuming Type I error = 0.05 and Type II error = 0.2 (80% power to detect this difference), then n=25 patients needed in each group.

      Study Design A prospective, randomised, double-blind controlled trial with participants masked to study arm (blocks will be performed under General Anaesthesia) and those involved in data collection also masked to the intervention. Patients will be asked to complete a questionnaire in the post operative period (QoR 15) which is a global assessment of the patients post operative recovery status. The QoR 15 scale is a validated means of assessing a patients quality of recovery. The questionnaire contains 15 questions and the mean+SD duration of time taken for patients to complete the questionnaire is 2.4+0.8 min.

      Treatment of study subjects Patients scheduled for Spinal Surgery will be screened for eligibility according to the criteria listed and eligible patients noted. These patients are admitted the day prior to surgery or morning of surgery when scheduled for an afternoon list. Eligible patients will be approached by an investigator and invited to give their consent to the study. They will be offered the Patient Information Leaflet (PIL) and the investigator will leave the patient for a minimum of ten minutes to consider. Patients who give written consent will be randomised to receive either ESB or No Block (control) after induction of general anaesthesia. Randomisation will be by table of random numbers, even numbers assigned ESB, odd numbers control. The designated group will then be written on a blank page and placed in a sealed envelope, which will be sequentially numbered, e.g. Patient Study Number 1 etc.

      Patients will be unconscious under GA when receiving either ESB , so will be masked to group allocation. Investigators collecting QoR-15 data will also be unaware of group allocation.

      All participants will have standard analgesia (Paracetamol, NSAIDS, Opiates) at the discretion of the treating Consultant Anaesthetist. 20mls 0.25% Levobupivicaine plus 2mg Dexamethasone will be used on each side in the ESP block.

      Patient characteristics and data will be prospectively recorded for 24 hr postoperatively. Intraoperative haemodynamic recordings and the use of rescue analgesia during the operation and in the recovery room will be taken from the Centricity Anaesthesia Information Management System an electronic recording system that has been in use in the Mater Anaesthesia department since 2016. Patients will complete QoR questionnaires manually on paper which will then be transferred into an electronic format. The questionnaires will be administered by Doctors or Nurses involved with the study. Patients will be asked to complete the questionnaire while they are in the recovery area after the operation and once they are fully awake.

      Inclusion Criteria Male and Female participants providing written informed consent, ASA grade 1- 4, age group 18 and over undergoing Posterior approach Spinal surgery involving 2 or more levels of decompression in the lumbar or thoracic regions.

      Exclusion Criteria Absence of informed written consent, pre existing infection at block site, severe coagulopathy, allergy to local anaesthesia, , previous history of opiate abuse, pre existing chronic pain condition, pre-existing dementia [because of need to co-operate in completing QoR-15 score day after surgery], decompression involving cervical levels of vertebrae

      Anticipated study start date

      1st August 2019 Anticipated study duration 6 months

      Safety Reporting Patients' routine medical care will continue during this clinical trial as per current practice. Both regional blocks are routinely used in our institution and therefore the health of participants will be monitored as it would be for all patients regardless of their participation in the trial. Adverse events will be recorded and managed along already existing local policies and guidelines.

      Statistics QoR and other variables will be compared between the groups using independent samples (unpaired) t-test for normally distributed continuous data and Mann-Whitney U test for non-parametric data

      Data Handling and record keeping Only the investigators will have access to the collated data. Data will be recorded initially on paper and then transcribed to electronic spreadsheet format, in coded format.

      Patients' names will not be recorded, study numbers assigned by randomisation will be recorded. This will allow follow up at 24 hours to assess block performance. The investigators will retain the "key" to identification. Data will be stored securely in the Department of Anaesthesia at the Mater Hospital, on a password-protected desktop computer stored in a locked office, such that only the investigators will have access.

      Electronically-recorded data will be secured by means of password protection/encryption. Data recorded on paper will be secured by lock and key

      Retention of essential documents The collated data collected by the investigators will be retained for 5 yr after analysis has completed. The original data in the patients' paper and electronic medical records will be unaffected.

      Quality Control and Quality assurance procedures ESP blocks are in routine use in our department currently. All Blocks will be performed by Anaesthesiologists with expertise in regional anaesthesia and who are familiar with the study. We will be following our local and international guidelines in terms of safe block performance. This would include appropriate monitoring of the patient as set out in the RA - UK guidelines, availability of resuscitation and airway equipment including the ready availability of Intra - lipid. All blocks will be performed by or supervised by experienced Anaesthesiologists using a validated in plane Ultrasound technique.

      Ethics There are no ethical issues regarding this study. Financing and Insurance/Indemnity All investigators will be MMUH staff covered by the clinical indemnity scheme [CIS]

      Clinical Study Report and publication policy Conclusions from the clinical trial, once complete, will be prepared for presentation at an academic meeting and for submission to an appropriate international, peer-reviewed journal

ELIGIBILITY:
Inclusion Criteria:Male and Female participants providing written informed consent, ASA grade 1- 4, age group 18 and over undergoing Posterior approach Spinal surgery involving 2 or more levels of decompression in the lumbar or thoracic regions.

-

Exclusion Criteria:Absence of informed written consent, pre existing infection at block site, severe coagulopathy, allergy to local anaesthesia, , previous history of opiate abuse, pre existing chronic pain condition, pre-existing dementia [because of need to co-operate in completing QoR-15 score day after surgery], decompression involving cervical levels of vertebrae, decompression due to queried or confirmed malignancy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-01-03 (Estimated)

PRIMARY OUTCOMES:
QoR 15 score | 24 hours post operatively
  a objective assessment of quality of recovery post surgery

SECONDARY OUTCOMES:
AUC of VRS Pain score versus time | 24 hours post op
  Area under the VRS pain score versus time
time to administration of first rescue analgesia after the block | 24 hours post op

CONTACTS AND LOCATIONS:
Overall Officials: Donal Buggy, MB Bch Bao, Principal Investigator — Professor of Anaesthesia and Perioperative Medicine
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Case report forms,
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Finnerty D, Ni Eochagain A, Ahmed M, Poynton A, Butler JS, Buggy DJ. A randomised trial of bilateral erector spinae plane block vs. no block for thoracolumbar decompressive spinal surgery. Anaesthesia. 2021 Nov;76(11):1499-1503. doi: 10.1111/anae.15488. Epub 2021 Apr 20. PMID 33878196
- [Derived] Finnerty DT, Buggy DJ. Efficacy of the erector spinae plane (ESP) block for quality of recovery in posterior thoraco-lumbar spinal decompression surgery: study protocol for a randomised controlled trial. Trials. 2021 Feb 17;22(1):150. doi: 10.1186/s13063-021-05101-2. PMID 33596968